CLINICAL TRIAL: NCT06185465
Title: Effectiveness and Safety of Using Prontosan Wound Irrigation Solution to Treat Bacterial Biofilm in Chronic Wound Patients With Secondary Infections: a Randomized, Controlled, Open Multicenter Study.
Brief Title: Effectiveness and Safety of Using Prontosan to Treat Bacterial Biofilm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Shenzhen Second People's Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-075
Record Dates: First submitted 2023-11-21; First posted 2023-12-29 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Irrigation Solution; Chronic Wound; Pressure Injury; Diabetic Foot Ulcer; Burns
Keywords: Prontosan wound irrigation solution; Prontosan; Chronic wound; Pressure Injury; Burns; Diabetic Foot Ulcer
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot; Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prontosan Wound Irrigation Solution rinse (Experimental): The test group is selected according to the randomization number of enrollment. For experimental group, Prontosan Wound Irrigation Solution is extracted with syringe (Dosage 1-2ml/cm2), and the wound is rinsed 1 cm from the wound. Then, Prontosan wound irrigation solution is used to saturate the gauze, and the gauze is applied to the wound for 15 minutes. After removing the gauze, cover it with oil gauze, then cover it with 8 layers of gauze and wrap it with a bandage.
  Interventions: Device: Prontosan Wound Irrigation Solution
- Normal Saline rinse (Active Comparator): For control group, Normal saline is extracted with syringe (Dosage 1-2ml/cm2), and the wound is rinsed 1 cm from the wound. Then, Normal saline is used to saturate the gauze, and the gauze is applied to the wound for 15 minutes. After removing the gauze, cover it with oil gauze, then cover it with 8 layers of gauze and wrap it with a bandage.
  Interventions: Device: Normal Saline

INTERVENTIONS:
Device: Prontosan Wound Irrigation Solution — After debridement surgery, the test group is selected according to the randomization number of enrollment. For experimental group, Prontosan Wound Irrigation Solution is extracted with syringe (Dosage 1-2ml/cm2), and the wound is rinsed 1 cm from the wound. Then, Prontosan wound irrigation solution is used to saturate the gauze, and the gauze is applied to the wound for 15 minutes. After removing the gauze, cover it with oil gauze, then cover it with 8 layers of gauze and wrap it with a bandage.
  Other Names: Debridement surgery
  Arms: Prontosan Wound Irrigation Solution rinse
Device: Normal Saline — After debridement surgery, the test group is selected according to the randomization number of enrollment. For control group, normal saline is extracted with syringe (Dosage 1-2ml/cm2), and the wound is rinsed 1 cm from the wound. Then, normal saline is used to saturate the gauze, and the gauze is applied to the wound for 15 minutes. After removing the gauze, cover it with oil gauze, then cover it with 8 layers of gauze and wrap it with a bandage.
  Other Names: Debridement surgery
  Arms: Normal Saline rinse

SUMMARY:
The goal of this prospective, multi-center, randomized, parallel-controlled, open-label clinical study is to evaluate the effectiveness and safety of Prontosan wound irrigation solution comparing with Normal Saline on the removal of wound bacterial biofilm through observing the morphological characteristics and development of bacterial biofilm in chronic wound patients with secondary infections. The main questions it aims to answer are:

* Difference in scoring the positive rate of bacterial biofilm before the first treatment and on the 7th day of treatment in Group A and Group B
* Difference in scoring the positive rate of bacterial biofilm before the first treatment and on the 3rd day of treatment in Group A and Group B .
* Positive detection rate of bacterial biofilm in group and group B before the first treatment, and on the 3rd and 7th day of treatment, and difference of the positive detection rate of biofilm among the two groups.
* 4-phase typing of bacterial biofilm detected in Group A, Group B and Group C before the first treatment, and on the 3rd and 7th day of treatment, and the proportion difference of 4-phase typing of biofilm among the two groups.
* Wound healing rate
* Skin Infection Rating Scale (SIRS) score.
* Distribution of inflammatory cells on the wound.
* Detection rate of bacteria/drug-resistant bacteria on the wound and their correlation with the detection rate of bacterial biofilm.

Participants will be randomized to experimental group or Control group, Prontosan Wound Irrigation Solution or normal saline will be extracted with syringe (Dosage 1-2ml/cm2), and the wound is rinsed 1 cm from the wound. Then, Prontosan wound irrigation solution or normal saline is used to saturate the gauze, and the gauze is applied to the wound for 15 minutes. After removing the gauze, cover it with oil gauze, then cover it with 8 layers of gauze and wrap it with a bandage.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign the informed consent form;
* 2. ≥18 years old;
* 3. Patients with chronic wound, eg. burns, and pressure injuries with stage 3 and 4. Diabetes foot ulcer with Wagner grade 2; (Staging and Wagner grading of stress injury can be found in attachments 1 and 2);
* 4. The length and width of a single wound in the wound area where the sampling point is located must be ≥2 cm, and the maximum length and width must be ≤10 cm;
* 5. The rapid smear test results of bacteria on the wound were positive;
* 6. The clinical symptoms of wound infection meet the following conditions: skin infection level scale score (SIRS) ≥ 8;
* 7. Patients identified by the investigator as having biofilm formation on the wound;
* 8. No eschar covering the wound surface.

Exclusion Criteria:

* 1. Patients administered with systemic antibiotics 48 hours before enrollment;
* 2. Patients with severe autoimmune diseases;
* 3. Patients with pressure injuries classified as Stage I and II; (Please refer to Attachment 1 for for pressure injury staging);
* 4. Diabetes foot ulcer with Wagner grade0- 1 and more than 3; (Wagner grading of stress injury can be found in attachments 2);
* 5. Female in pregnancy or lactation period;
* 6. Those who have participated in clinical trials of drugs or devices within one month before the first treatment;
* 7. Patients who are allergic to any component of the research device;
* 8. Those who are currently using tumor chemotherapy drugs during screening;
* 9. Any condition that, in the opinion of the investigator, may increase the risk to the subjects or otherwise affect the evaluation of efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-02-21 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Difference in scoring the positive rate of bacterial biofilm before the first treatment and on the 7th day of treatment in Group A and Group B | Day0, Day7
  Difference in scoring the positive rate of bacterial biofilm=the total score of 3 tissues before treatment- the total score of 3 tissues treatment after 7days. To compare the score difference between 2 groups after the difference is calculated.

SECONDARY OUTCOMES:
Difference in scoring the positive rate of bacterial biofilm before the first treatment and on the 3rd day of treatment in Group A and Group B | Day0, Day3
  Difference in scoring the positive rate of bacterial biofilm=the total score of 3 tissues before treatment- the total score of 3 tissues treatment after 3 days. To compare the score difference between 2 groups after the difference is calculated
Positive detection rate of bacterial biofilm in group and group B before the first treatment, and on the 3rd and 7th day of treatment, and difference of the positive detection rate of biofilm among the two groups | Day0, Day3,Day7
  If any of the 3 samples is tested positive for the biofilm, the result will be judged positive (+); If no biofilm is detected in the 3 samples, the result will be judged negative (-).
4-phase typing of bacterial biofilm detected in Group A, Group B and Group C before the first treatment, and on the 3rd and 7th day of treatment, and the proportion difference of 4-phase typing of biofilm among the two groups | Day0, Day3,Day7
  Typing I: 0 point is scored in case of free bacteria, i.e., dispersed phase of monomer bacteria; Typing II: 0 points are scored in case of bacterial adhesion, i.e., aggregation phase of monomer bacteria; Typing III&IV: 3 points are scored in case of mature bacterial biofilm, i.e., closed phase of colony bacteria; 3 points are scored in case of spreading of bacterial biofilm, i.e., open phase of colony bacteria.
Wound healing rate | Day0, Day3,Day7
  The wound is covered with sterile mesh film before the first treatment, and on the 3rd and 7th day of treatment, the wound area is measured and recorded, and the difference in wound healing rate among the two groups is compared.
Skin Infection Rating Scale (SIRS) score | Day0, Day3,Day7
  o Skin Infection Rating Scale (SIRS) scoring is conducted and recorded before the first treatment, and on the 3rd and 7th day of treatment to compare the differences of SIRS scores among the two groups.
  SIRS scoring Items include Exudate / pus, Scabbing, Erythema/Inflammation, Tissue edema, Tissue fever, Pruritus and Pain. The scores of every items are 0=none, 1=mild, 2= Moderate, 3= severe.
Distribution of inflammatory cells on the wound | Day0, Day3,Day7
  The H-E staining pathological sections of inflammatory cells on the wound are carried out before the first treatment, and on the 3rd and 7th day of treatment to compare the differences in the distribution type (Monocytes/Neutrophils/Lymphocytes) and quantity(No infiltration, mild infiltration, moderate infiltration, severe infiltration) of inflammatory cells on the wound among the two groups.
  mild infiltration refers to the infiltration of less than or equal to 10 inflammatory cells； moderate infiltration refers to the infiltration of 11-50 inflammatory cells; severe infiltration refers to the infiltration of more than 50 inflammatory cells.
Detection rate of bacteria/drug-resistant bacteria on the wound and their correlation with the detection rate of bacterial biofilm | Day0, Day3,Day7
  According to the test results, the number of bacteria positive cases and number of drug-resistant positive bacteria cases are counted, and the difference in anti-infection ability of the two groups after 3 and 7 days of wound treatment is compared by the number of positive cases/total number of burn patients in each group and the number of drug-resistant bacteria positive cases/total number of burn patients in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Jia'ao Yu, Professor, Study Chair — The First Hospital of Jilin University; Jun Wu, Professor, Principal Investigator — Shenzhen Second People's Hospital; Zhaohong Chen, Professor, Principal Investigator — Fujian Medical University Union Hospital
Locations (3):
- China (3):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - First Hospital of Jilin University, Changchun, Jilin
  - Shenzhen Second People's Hospital, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No
Not share.